CLINICAL TRIAL: NCT05807516
Title: Study of the Impact of Neoadjuvant Therapy on the Heterogeneity of Triple Negative Breast Cancer Through Single-cell RNA Sequencing (scRNAseq) and Whole-exome Sequencing (WES)
Brief Title: Single-cell RNAseq Breast Cancer
Acronym: SCRBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1637/21
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Single-Cell Gene Expression Analysis; Exome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Single-cell RNA sequencing (scRNAseq), whole-exome sequencing (WES) — Combined both retrospective and prospective observational design

SUMMARY:
Molecular characterization of persistent tumor cells remaining after NAC and infiltrating immune cells, for example, M2 macrophages, could strongly contribute to identifying targeted therapeutic approaches for this disease.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) represents approximately 15-20% of all breast cancers. Its features are lack of expression of estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (Her2). TNBC exhibits a biologically aggressive behavior and a high inter- and intra-tumor molecular heterogeneity which has recently been highlighted also in single cell RNAseq (scRNAseq) studies. Patients with TNBC often have less positive outcomes then other breast cancer subtypes, due to the absence of specific therapeutic targets.

Results of single cell RNA sequencing (scRNAseq) in TNBC before and after treatment with chemotherapy (NAC) were recently reported for a small group of patients. Genetic alterations are also investigated by Whole Exome Sequencing (WES).

In addition scRNAseq analysis confirmed the presence of a high percentage of M2 macrophages in TNBC and tumor-adjacent tissue. These macrophages are clinically relevant and able to predict outcome in TNBC.

Based on the above evidence, we hypothesize that molecular characterization of persistent tumor cells remaining after NAC and infiltrating immune cells, for example, M2 macrophages, could strongly contribute to identifying targeted therapeutic approaches for this disease.

We will conduct a pilot study with a combined retrospective and prospective observational design.

Cancer patients diagnosed with histologically proven primary invasive breast cancer with a stage IIA to IIIB and assessed at the molecular level and defined as TNBC, will be eligible to participate to the study. Furthermore, only patients with a tumor >1.5cm in size will be considered, which is the selection criterion for the administration of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven primary invasive breast cancer >1.5cm in size, with molecular assessed stage IIA to IIIB defined as TNBC, and who will undergo neoadjuvant chemotherapy and subsequent surgery (and/or have undergone - retrospective part).
* informed consent (prospective part)

Exclusion Criteria:

* pregnancy, metastatic breast cancer, previous chemotherapy, hormone therapy, radiation therapy, previous other cancers or contralateral breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The retrospective study will be performed using only formalin-fixed paraffin-embedded (FFPE) tissue samples for protein expression profiling (proteomics) from patients withthe above inclusion/exclusion criteria from the archives of the Pathological anatomy of the IRE.
  The prospective study foresees the collection of biological samples by the centers involved in the study and the freezing of all the samples at the IRE Biological Bank.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate chemoterapy effect | 26 months
  Decipher, through the execution of scRNAseq profiles, the transcriptional reprogramming that occurs during chemotherapy (NAC) in triple negative breast cancers (TNBC) and provide information of prognostic and/or predictive relevance of response to NAC

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Policlinico Umberto I, Roma
  - "Regina Elena" National Cancer Institute, Rome

IPD SHARING:
Plan to Share IPD: Undecided